CLINICAL TRIAL: NCT03549910
Title: A Multicenter, Random Control Study: Early Use of Airway Pressure Release Ventilation Updated (APRVplus) Protocol in Acute Respiratory Disease Syndrome (ARDS)
Brief Title: A Multicenter, Random Control Study :Early Use of Airway Pressure Release Ventilation (APRVplus) Protocol in ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, Director of department of Critical Care Medicine, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Huaxi ICU-APRV
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early use of APRVplus protocol in ARDS (Experimental): physiology-driven APRVplus protocol
  Interventions: Procedure: APRVplus protocol
- Low tidal volume ventilation (Other): Low tidal volume lung protective ventilation
  Interventions: Procedure: Low tidal volume ventilation

INTERVENTIONS:
Procedure: APRVplus protocol — Physiology-driven APRVplus protocol
  Arms: Early use of APRVplus protocol in ARDS
Procedure: Low tidal volume ventilation — Low tidal volume lung protective ventilation
  Arms: Low tidal volume ventilation

SUMMARY:
Animal experimentals have shown that the more physiology-driven airway pressure release ventilation (APRV) methodologies in ARDS may significantly improve alveolar recruitment and gas exchange, increased homogeneity, and attenuate lung injury, without circulatory depression, as compared with conventional low tial volume lung protective ventilation. our previous single centre,random control study showed that clinical benefit for early use of APRV in ARDS. Nonetheless, clinical data on ARDS are still limited, most of them derived from small clinical trials in which variable outdated APRV settings were used, consequently, the findings of these studies were controversial.

Additionally, the previous single-centre,random control study showed that clinical benefit for APRV.Therefore,the investigators are ready to design a multiple centres,random control study to further verify the effect of APRV plus protocol in ARDS.

DETAILED DESCRIPTION:
All the patients included will be randomly assigned to receiving APRV plus protocol or low tidal volume ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and severe acute respiratory distress syndrome,according to the Berlin definition of ARDS
* receiving tracheal intubation and mechanical ventilation was no longer than 48 hours

Exclusion Criteria:

* Pregnancy
* The expected duration of mechanical ventilation was less than 48 hours
* Intracranial hypertension (suspected or confirmed)
* Neuromuscular disorders that are known to prolong the need for mechanical ventilation
* Known or suspected chronic obstructive pulmonary disease(COPD)
* Terminal stage of disease
* Pneumothorax (drained or not)at enrollment
* Treatment with extracorporeal support (ECMO) at enrollment
* There was a lack of commitment to life support.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
mortality | Day 28
  mortality at Day28

SECONDARY OUTCOMES:
Mechanical ventilation free days | Day 28
  Mechanical ventilation free days at Day28
oxygenation | from enrollment to Day7
  oxygenation index:PaO2:fiO2
repiratory system compliance | from enrollment to Day7
  static repiratory system compliance (ml/cmH2O)
MAP | during the mechanical ventilation procedure
  mean arterial pressure
sedation depth | during the mechanical ventilation procedure
  RASS scores
Sedative drug | during the mechanical ventilation procedure
  the total dose of Sedative drug
successful extubation rate | during the mechanical ventilation procedure
  the rate of successful extubation

OTHER OUTCOMES:
adverse events related to mechanical ventilation | during the mechanical ventilation procedure
  including pneumothorax,VAP,and so on

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yan, Study Chair — Department of Critical Care Medicine
Locations (1):
- West China Hospital,Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou Y, Cheng J, Zhu S, Dong M, Lv Y, Jing X, Kang Y. Early pathophysiology-driven airway pressure release ventilation versus low tidal volume ventilation strategy for patients with moderate-severe ARDS: study protocol for a randomized, multicenter, controlled trial. BMC Pulm Med. 2024 May 23;24(1):252. doi: 10.1186/s12890-024-03065-y. PMID 38783268